CLINICAL TRIAL: NCT05293639
Title: Assessment of Safety and Effectiveness in Treatment Management of Atrial Fibrillation With the BWI IRE Ablation System (AdmIRE)
Brief Title: Assessment of Safety and Effectiveness in Treatment Management of Atrial Fibrillation With the BWI IRE Ablation System
Acronym: AdmIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BWI201910
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Results first posted 2025-04-04 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation
Keywords: Interventional; Irreversible electroporation; Paroxysmal atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Irreversible Electroporation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment Group (Experimental): PFA ablation using a circular multi-electrode pulsed electrical field catheter and multichannel generator
  Interventions: Device: Pulse Field Ablation

INTERVENTIONS:
Device: Pulse Field Ablation — PFA ablation using a circular multi-electrode pulsed electrical field catheter and multichannel generator

SUMMARY:
To demonstrate the safety and 12-month effectiveness of the VARIPULSE™ Catheter when used in conjunction with the TRUPULSE™ Generator for pulmonary vein isolation (PVI) in the treatment of subjects with symptomatic paroxysmal atrial fibrillation.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, multi-center, clinical evaluation of the Biosense Webster IRE Ablation system to demonstrate safety and long-term effectiveness for the treatment of drug refractory symptomatic PAF. The BWI IRE Ablation System consists of the VARIPULSE™ Catheter and TRUPULSE™ Generator. In conjunction with CARTO™ 3 system, it is indicated for PVI of patients with drug refractory paroxysmal atrial fibrillation.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosed with Symptomatic Paroxysmal Atrial Fibrillation with

  1. At least two symptomatic AF episodes within last six months from enrollment.
  2. At least one ectrocardiographically documented AF episode within twelve (12) months prior to enrollment.
* Failed at least one Class I or Class III antiarrhythmic drug.

Exclusion Criteria:

* Previously diagnosed with persistent AF (> 7 days in duration).
* AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause.
* Previous surgical or catheter ablation for AF.
* Patients known to require ablation outside the PV region
* Documented severe dilatation of the LA (LAD >50mm) antero-posterior diameter on imaging within 6 months prior to enrollment.
* Documented LA thrombus by imaging within 48 hours of the procedure.
* Documented severely compromised LVEF (<40%) by imaging within 6 months prior to enrollment
* Uncontrolled heart failure or New York Heart Association Class III or IV
* History of blood clotting, bleeding abnormalities or contraindication to anticoagulation (heparin, warfarin, or dabigatran),
* Documented thromboembolic event (including TIA) within the past 12 months
* Previous PCI/MI within the past 2 months
* Coronary Artery Bypass Grafting (CABG) surgery within the past 6 months (180 days)
* Valvular cardiac surgical/percutaneous procedure
* Unstable angina within 6 months
* Anticipated cardiac transplantation, cardiac surgery, or other major surgery within the next 12 months.
* Significant pulmonary disease or any other disease or malfunction of the lungs or respiratory system that produces severe chronic symptoms.
* Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment in this study
* Prior diagnosis of pulmonary vein stenosis
* Pre-existing hemi diaphragmatic paralysis
* Acute illness, active systemic infection, or sepsis
* Presence of intracardiac thrombus, myxoma, tumor, interatrial baffle or patch or other abnormality that precludes catheter introduction or manipulation.
* Severe mitral regurgitation
* Presence of implanted pacemaker or Implantable Cardioverter-Defibrillator (ICD) or other implanted metal cardiac device that may interfere with the IRE energy field.
* Presence of a condition that precludes vascular access
* Current enrollment in an investigational study evaluating another device or drug.
* Women who are pregnant, lactating, or who are of child-bearing age and plan on becoming pregnant during the course of the clinical investigation.
* Life expectancy less than 12 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Biosense Webster Inc. Clinical Trial, Study Director — Biosense Webster, Inc.
Locations (30):
- United States (30):
  - Grandview Medical Center, Birmingham, Alabama
  - Phoenix Cardiovascular Research, Phoenix, Arizona
  - Arrhythmia Research Group (St. Bernards), Jonesboro, Arkansas
  - Cardiovascular Group of Marin/SF Med Group, Larkspur, California
  - Hoag Memorial Hospital, Newport Beach, California
  - San Diego Cardiac Center, San Diego, California
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Florida Hospital, Orlando, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Evanston Hospital / Northshore, Evanston, Illinois
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Morristown Medical Center, Morristown, New Jersey
  - South Shore University Hospital, Bay Shore, New York
  - New York University Langone Med Center, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Wakemed Heart and Vascular, Raleigh, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Baylor Research Institute, Plano, Texas
  - Inova Fairfax Medical Center, Falls Church, Virginia
  - Virginia Commonwealth Uninversity, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Devices Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

REFERENCES:
- [Derived] Di Biase L, Reddy VY, Bahu M, Newton D, Liu CF, Sauer WH, Goyal S, Iyer V, Nair D, Osorio J, Mansour M, Calkins H, Wazni O, Natale A. Early versus late atrial fibrillation recurrence after pulsed field ablation: insights from the admIRE trial. Europace. 2025 Feb 5;27(2):euaf007. doi: 10.1093/europace/euaf007. PMID 39820338
- [Derived] Reddy VY, Calkins H, Mansour M, Wazni O, Di Biase L, Bahu M, Newton D, Liu CF, Sauer WH, Goyal S, Iyer V, Nair D, Athill C, Hussein A, Whalen P, Melby D, Natale A; AdmIRE Trial Investigators. Pulsed Field Ablation to Treat Paroxysmal Atrial Fibrillation: Safety and Effectiveness in the AdmIRE Pivotal Trial. Circulation. 2024 Oct 8;150(15):1174-1186. doi: 10.1161/CIRCULATIONAHA.124.070333. Epub 2024 Sep 11. PMID 39258362

RESULTS

PARTICIPANT FLOW:
Groups:
- Pilot Safety Analysis Set: Participants enrolled in the pilot phase with symptomatic paroxysmal atrial fibrillation (PAF) and had an insertion of the Biosense Incorporated Webster (BWI) Irreversible Electroporation (IRE) Ablation System (with or without delivery of PFA), underwent electrophysiology mapping and pulsed field ablation (PFA) for treatment of Antiarrhythmic Drug (AAD) refractory symptomatic PAF.
- Pivotal Roll-In Analysis Set: Participants enrolled in the pivotal roll-In phase with symptomatic paroxysmal atrial fibrillation (PAF) had an insertion of the BWI IRE Ablation System and PFA delivery, underwent electrophysiology mapping and PFA for treatment of AAD refractory symptomatic PAF.
- Pivotal Main Safety Analysis Set: Participants enrolled in the in pivotal main phase with symptomatic PAF had an insertion of the BWI IRE Ablation System (with or without delivery of PFA), underwent electrophysiology mapping and PFA for treatment of AAD refractory symptomatic PAF.
Period: Overall Study
Arm/Group | Pilot Safety Analysis Set | Pivotal Roll-In Analysis Set | Pivotal Main Safety Analysis Set
Started | 21 | 64 | 277
Completed | 20 | 62 | 269
Not Completed | 1 | 2 | 8
Not completed — Withdrawal by Subject | 1 | 1 | 2
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 5
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pilot Safety Analysis Set | Pivotal Roll-In Analysis Set | Pivotal Main Safety Analysis Set | Total
Number analyzed (Participants) | 21 | 64 | 277 | 362
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age (Year) | 62.1 (10.20) | 61.2 (8.97) | 61.5 (10.30) | 61.5 (10.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 26 | 99 | 134
  Male | 12 | 38 | 178 | 228
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 7 | 8
  Not Hispanic or Latino | 20 | 57 | 215 | 292
  Unknown or Not Reported | 1 | 6 | 55 | 62
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 4 | 5
  Asian | 0 | 3 | 12 | 15
  Black or African American | 1 | 3 | 7 | 11
  White | 20 | 54 | 228 | 302
  Other | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 3 | 25 | 28

OUTCOME MEASURES:

1. Primary Outcome: Pivotal Main Phase Modified Intent-To-Treat (mITT) Analysis Set: Number of Participants With Primary Adverse Events (PAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. PAEs included the following AEs: Phrenic Nerve Paralysis (permanent), Stroke/Cerebrovascular accident (CVA), Major Vascular Access Complication/Bleeding, Thromboembolism, Myocardial Infarction, Transient Ischemic Attack (TIA), Pericarditis, Pulmonary Edema (Respiratory Insufficiency), Heart Block, and Vagal Nerve Injury/ Gastroparesis.
Time Frame: From Day 0 to Day 7 post catheter insertion on Day 0
Population: mITT analysis set included all participants enrolled in the pivotal main phase who met eligibility criteria and had insertion of the study catheter. Here, "N" (Overall number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Pivotal Main Phase mITT Analysis Set: Participants enrolled in the in pivotal main phase with symptomatic PAF had an insertion of the BWI IRE Ablation System (with or without delivery of PFA), underwent electrophysiology mapping and PFA for treatment of AAD refractory symptomatic PAF.
Arm/Group | Pivotal Main Phase mITT Analysis Set
Number analyzed (Participants) | 272
Participants | 8

2. Primary Outcome: Pilot Safety Analysis Set and Pivotal Roll-In Analysis Set: Number of Participants With Primary Adverse Events (PAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. PAEs included the following AEs: Phrenic Nerve Paralysis (permanent), Stroke/CVA, Major Vascular Access Complication/Bleeding, Thromboembolism, Myocardial Infarction, Transient Ischemic Attack (TIA), Pericarditis, Pulmonary Edema (Respiratory Insufficiency), Heart Block, and Vagal Nerve Injury/ Gastroparesis.
Time Frame: From Day 0 to Day 7 post catheter insertion on Day 0
Population: Pilot phase used the safety analysis set, included participants enrolled in the Pilot phase and had insertion of the study catheter (with or without delivery of PFA). Pivotal roll-In phase analysis set included all participants enrolled and had insertion of the study catheter and undergone PFA delivery with the IRE ablation system. Here, "N" (Overall number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Pivotal Roll-In Analysis Set: Participants enrolled in the pivotal roll-In phase with symptomatic paroxysmal atrial fibrillation (PAF) had an insertion of the Biosense Webster (BWI) Irreversible Electroporation (IRE) Ablation System and PFA delivery, underwent electrophysiology mapping and pulsed field ablation (PFA) for treatment of Antiarrhythmic Drug (AAD) refractory symptomatic paroxysmal AF.
Arm/Group | Pilot Safety Analysis Set | Pivotal Roll-In Analysis Set
Number analyzed (Participants) | 20 | 63
Participants | 0 | 0

3. Primary Outcome: Pivotal Main Phase Per-Protocol (PP) Analysis Set: Number of Participants With Freedom of Documented Atrial Tachyarrhythmia
Description: Number of Participants With freedom from documented (symptomatic and asymptomatic) atrial tachyarrhythmia (atrial fibrillation [AF], atrial tachycardia [AT], or atrial flutter [AFL] of unknown origin positive) episodes based on electrocardiographic data (greater than or equal to [>=] 30 seconds on an electrocardiogram [ECG], sponsor-provided cardiac event monitor [CEM], or Holter device) during the effectiveness evaluation period (Day 91-365 post catheter insertion procedure) and freedom from the following failure modes: acute procedural failure, repeat ablation failure, non-study catheter failure, AAD failure, continuous AF/AT/AFL of unknown origin on ECG, any Direct Current Cardioversion (DCCV) procedure were reported.
Time Frame: Day 91 to Day 365 post catheter insertion on Day 0
Population: PP analysis set included all participants enrolled in the pivotal main phase who were treated for the study-related arrhythmia with the study catheter and without protocol deviations that would affect the scientific integrity of the study. Here "N" (Overall number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Pivotal Main Phase PP Analysis Set: Participants enrolled in the in pivotal main phase with symptomatic PAF had an insertion of the BWI IRE Ablation System (with or without delivery of PFA), underwent electrophysiology mapping and PFA for treatment of AAD refractory symptomatic PAF.
Arm/Group | Pivotal Main Phase PP Analysis Set
Number analyzed (Participants) | 246
Participants | 183

4. Primary Outcome: Pilot Safety Analysis Set and Pivotal Roll-In Analysis Set: Number of Participants With Freedom of Documented Atrial Tachyarrhythmia
Description: Number of Participants With freedom from documented (symptomatic and asymptomatic) atrial tachyarrhythmia (AF, AT, or AFL of unknown origin positive) episodes based on electrocardiographic data (>=30 seconds on an ECG, CEM, or Holter device) during the effectiveness evaluation period (Day 91-365 post catheter insertion) and freedom from the following failure modes: acute procedural failure, repeat ablation failure, non-study catheter failure, AAD failure, continuous AF/AT/AFL of unknown origin on ECG, any DCCV procedure were reported.
Time Frame: Day 91 to Day 365 post catheter insertion on Day 0
Population: Pilot phase used the safety analysis set, included participants enrolled in the Pilot phase and had insertion of the study catheter (with or without delivery of PFA). Pivotal roll-In phase analysis set included all participants enrolled and had insertion of the study catheter and undergone PFA delivery with the IRE ablation system. Here "N" (Overall number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Safety Analysis Set | Pivotal Roll-In Analysis Set
Number analyzed (Participants) | 20 | 63
Participants | 16 | 43

5. Secondary Outcome: Pivotal Main Phase PP Analysis Set: Change From Baseline in Overall Atrial Fibrillation Effect on Quality-of-Life Questionnaire (AFEQT) Total Score
Description: Change from baseline in overall AFEQT total score were reported. Change in the AFEQT score included 20 questions on a 7-point Likert scale. Questions 1-18 evaluated Health Related Quality of Life (HRQoL) and questions 19-20 were related to the patient's satisfaction with treatment. The first 18 questions were used to calculate the overall AFEQT score. The total AFEQT scores was calculated as 100 minus ([Sum of severity for all questions answered minus number of questions answered) divided by total number of questions answered*6])*100. The overall AFEQT scores ranged from 0 (complete disability) to 100 (no disability). Therefore, a positive change in score corresponded to improvement in QoL.
Time Frame: Baseline, and 12 months post catheter insertion on Day 0
Population: PP analysis aet included all participants enrolled in the pivotal main phase who were treated for the study-related arrhythmia with the study catheter and without protocol deviations that would affect the scientific integrity of the study. Here "N" (Overall number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pivotal Main Phase PP Analysis Set
Number analyzed (Participants) | 239
score on a scale | 32.03 (23.075)

6. Secondary Outcome: Pilot Safety Analysis Set and Pivotal Roll-In Analysis Set: Change From Baseline in Overall Atrial Fibrillation Effect on Quality-of-Life Questionnaire (AFEQT) Total Score
Description: Change from baseline in overall AFEQT total score were reported. Change in the AFEQT score included 20 questions on a 7-point Likert scale. Questions 1-18 evaluated HRQoL and questions 19-20 were related to the patient's satisfaction with treatment. The first 18 questions were used to calculate the overall AFEQT score. The total AFEQT scores was calculated as 100 minus ([Sum of severity for all questions answered minus number of questions answered) divided by total number of questions answered*6])*100. The overall AFEQT scores ranged from 0 (complete disability) to 100 (no disability). Therefore, a positive change in score corresponded to improvement in QoL.
Time Frame: Baseline, and 12 months post catheter insertion on Day 0
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pilot Safety Analysis Set | Pivotal Roll-In Analysis Set
Number analyzed (Participants) | 20 | 62
score on a scale | 31.13 (27.150) | 34.98 (24.553)

ADVERSE EVENTS:
Time Frame: From screening up to 12 months
Description: Adverse Events from enrollment through study exit were reported. SAE and NSAE presented below include PAE and all-cause mortality events.
Arm/Group | Pilot Safety Analysis Set | Pivotal Roll-In Analysis Set | Pivotal Main Safety Analysis Set
All-Cause Mortality (participants affected / at risk) | 0/21 | 1/64 | 0/277
Serious Adverse Events (participants affected / at risk) | 2/21 | 7/64 | 31/277
Other Adverse Events (participants affected / at risk) | 12/21 | 23/64 | 109/277
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pilot Safety Analysis Set (N=21) | Pivotal Roll-In Analysis Set (N=64) | Pivotal Main Safety Analysis Set (N=277)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pilot Safety Analysis Set (N=21) | Pivotal Roll-In Analysis Set (N=64) | Pivotal Main Safety Analysis Set (N=277)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercoagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1) | 8 (9)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Sinus arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Dermoid cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 5 (5)
Vitreous detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 3 (3)
Chest pain (General disorders) | 0 (0) | 1 (1) | 2 (2)
Fatigue (General disorders) | 0 (0) | 3 (3) | 1 (1)
Hernia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (3)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
COVID-19 (Infections and infestations) | 0 (0) | 5 (5) | 16 (16)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Groin infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (3)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Tinea cruris (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abdominal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Incision site complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (3)
Splinter (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Vascular access site bruising (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Vascular access site inflammation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Palate injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Bleeding time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QRS complex prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram change (Investigations) | 0 (0) | 0 (0) | 1 (1)
Prostatic specific antigen increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Femoral bruit (Investigations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Ankle deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Aura (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ophthalmic migraine (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Vocal cord paresis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Migraine with aura (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Device breakage (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Bladder dilatation (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 6 (7)
Adnexa uteri cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Haematospermia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myxoid cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Fibromuscular dysplasia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 4 (4)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT05293639/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT05293639/SAP_002.pdf